CLINICAL TRIAL: NCT03290352
Title: Pretreatment Quality of Life as a Predictor of Distant Metastasis-Free Survival and Overall Survival in Patients With Head and Neck Cancer Who Underwent Free Flap Reconstruction
Brief Title: Pretreatment Quality of Life as a Predictor of Distant Metastasis-Free Survival and Overall Survival in Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Chia-Chin Lin, Professor, Taipei Medical University
Other Study IDs: HKU_1
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and neck cancer patients: Patients with oral cavity, tongue, gingival, pharyngeal, laryngeal, or salivary gland cancer and cervical lymph node metastasis who received free flap reconstruction would be enrolled in this study. However, we excluded the patients with distant metastasis identified in their medical records, and those undergoing reconstruction other than anterolateral thigh, fibular bone and radial forearm flaps.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients who enrolled in the study were asked to respond to the University of Washington Quality of Life Questionnaire one week before undergoing free flap reconstruction.

SUMMARY:
This study shed light on an under-researched area by examining the prognostic associations of pre-treatment QoL with overall survival and distant metastasis free survival among patients with head and neck cancer who underwent free flap reconstruction. In addition, a validated instrument specific to head and neck cancer, i.e. the University of Washington Quality of Life Questionnaire (UW-QoL) was adopted.

DETAILED DESCRIPTION:
The importance of patient-related outcomes, especially quality of life (QoL) has been recently emphasized in the field of oncology. In conjunction with traditional biomedical indicators, QoL is recognized as a reliable parameter to reflect the health status of patients with malignancy. A growing body of evidence even points out that QoL can produce prognostic information which goes beyond biomedical indicators. In particular, since QoL may decline before any possible deterioration in health can be detected by existing biomedical measures, assessing pre-treatment QoL possibly helps identify the patients who are susceptible to a higher risk of mortality after they receive cancer treatment, which may greatly facilitate the process of clinical decision making. Despite the importance of pre-treatment QoL, its prognostic associations with overall survival and distant metastasis free survival still remain relatively under-explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oral cavity, tongue, gingival, pharyngeal, laryngeal, or salivary gland cancer and cervical lymph node metastasis, and
* Received free flap reconstruction between November 2010 and June 2014 at a medical university hospital

Exclusion Criteria:

* Patients with distant metastasis identified in their medical records, or
* Undergoing reconstruction other than anterolateral thigh, fibular bone and radial forearm flaps

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Head and neck cancer patients undergoing free-flap reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Overall survival of head and neck cancer patients with free-flap reconstruction | 3 years 8 months

SECONDARY OUTCOMES:
Distant metastasis free survival of head and neck cancer patients with free-flap reconstruction | 3 years 8 months

IPD SHARING:
Plan to Share IPD: Undecided